CLINICAL TRIAL: NCT01234428
Title: Esophageal Dysmotility Disorders Following Laparoscopic Gastric Banding - An Underestimated Complication.
Brief Title: Esophageal Dysmotility and Dilatation After Laparoscopic Gastric Banding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spital STS AG (Industry)
Collaborators: Department of Medicine, Spital STS AG Thun (Unknown)
Responsible Party: Markus Naef, MD, MBA, Department of Surgery, Spital STS AG Thun, Switzerland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOB-12-STS-AG
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-11

CONDITIONS: Esophageal Motility Disorders
Keywords: laparoscopy; adjustable gastric banding; morbid obesity; esophageal motility; esophageal dilatation
MeSH Terms: conditions — Esophageal Motility Disorders; Obesity, Morbid | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- surgery (Other)
  Interventions: Procedure: Laparoscopic surgery; Procedure: gastric banding

INTERVENTIONS:
Procedure: Laparoscopic surgery — Gastric banding
Procedure: gastric banding — laparoscopic gastric banding
  Other Names: morbid obesity

SUMMARY:
The purpose of this study is to determine whether esophageal dysmotility and dilatation is an important complication in the long term follow-up following laparoscopic gastric banding for morbid obesity.

DETAILED DESCRIPTION:
Using a yearly barium swallow the diameter of the esophagus will be monitored over the period.

ELIGIBILITY:
Inclusion Criteria:

* BMI more than 40

Exclusion Criteria:

* BMI below 40

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 1998-06; Primary Completion 2009-06 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
esophageal dilatation | yearly follow-up over 12 year period
  esophageal dilatation or dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Markus Naef, MD, MBA, Principal Investigator — Spital STS AG Thun, Switzerland
Locations (1):
- Department of Surgery, Spital STS AG Thun, Thun, Switzerland

REFERENCES:
- [Derived] Naef M, Mouton WG, Naef U, van der Weg B, Maddern GJ, Wagner HE. Esophageal dysmotility disorders after laparoscopic gastric banding--an underestimated complication. Ann Surg. 2011 Feb;253(2):285-90. doi: 10.1097/SLA.0b013e318206843e. PMID 21169806